CLINICAL TRIAL: NCT03178864
Title: Multicentre, Prospective Randomized Open Label, Blinded-endpoint (PROBE) Controlled Trial of Early Anticoagulation With Rivaroxaban Versus Standard of Care in Determining Safety at 365 Days in Symptomatic Cerebral Venous Thrombosis
Brief Title: Study of Rivaroxaban for CeREbral Venous Thrombosis
Acronym: SECRET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Thalia Field, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17-00440
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Venous Thrombosis
Keywords: cerebral venous thrombosis; anticoagulation
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Rivaroxaban; Standard of Care; Heparin; Warfarin; Dalteparin; Enoxaparin; Tinzaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban
  Interventions: Drug: Rivaroxaban
- Standard of care (Active Comparator): Unfractionated heparin Low-molecular weight heparin (dalteparin, enoxaparin, tinzaparin) Warfarin
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 20 mg daily (15 mg daily in participants with a CrCl 30-49 mL/min as per the Cockroft-Gault equation)
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Standard of care — Accepted standard of care as per American Heart Association/American Stroke Association Guidelines (initial use of unfractionated heparin or low-molecular weight heparin with transition to an oral vitamin K antagonist or continuation with low-molecular weight heparin) with choice of agent at the treating physician's discretion.
  Other Names: Heparin, Coumadin, Fragmin, Lovenox, Innohep
  Arms: Standard of care

SUMMARY:
SECRET examines the safety of rivaroxaban versus standard-of-care for treatment of symptomatic cerebral venous thrombosis, initiated within 14 days of diagnosis.

DETAILED DESCRIPTION:
SECRET is an open-label, randomized, controlled, phase II study that will assess the safety of rivaroxaban, a non-vitamin K antagonist oral anticoagulant (NOAC), compared with standard-of-care (unfractionated or low-molecular weight heparin with transition to warfarin [INR 2.0-3.0], or continued low molecular-weight heparin) for cerebral venous thrombosis. Recruitment will occur at 17 high-volume stroke research centres across Canada over 3 years. During the pilot phase, 50 adult patients within 14 days of symptomatic cerebral venous thrombosis diagnosis will be randomized to receive rivaroxaban 20 mg daily versus standard of care (warfarin or low-molecular weight heparin). Patients will be followed for 1 year. The feasibility of recruitment will be tested during the pilot phase and outcomes refined for a future Phase III trial.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18 and above
2. New diagnosis of symptomatic cerebral venous thrombosis as confirmed on CT venogram or MR venogram
3. Ability to randomize within 14 days of neuroimaging-confirmed diagnosis
4. The treating clinician is of the opinion that the patient is appropriate for oral anticoagulation as per standard of care
5. Patient or legally authorized representative is able to give written informed consent

Exclusion criteria:

1. Patient has known antiphospholipid antibody syndrome (APLS; lupus anticoagulant, anti-beta 2-glycoprotein I antibodies, and anticardiolipin antibody) by Sapporo-Sydney criteria with a previous history of venous or arterial thrombosis
2. Patient is anticipated to require invasive procedure (e.g. lumbar puncture, thrombectomy, hemicraniectomy) prior to initiation of oral anticoagulation**
3. Patient is unable to swallow due to depressed level of consciousness†
4. Impaired renal function (i.e., CrCl < 30 mL/min using Cockroft-Gault equation)
5. Pregnancy; if a woman is of childbearing potential a urine or serum beta human chorionic gonadotropin (β-hCG) test is positive
6. Breastfeeding at the time of randomization
7. Bleeding diathesis or other contraindication to anticoagulation
8. Any concurrent medical condition requiring mandatory antiplatelet or anticoagulant use
9. Concomitant use of strong CYP3A4 inducers (e.g., ongoing use of dilantin, carbamazepine, HIV protease inhibitors) or CYP3A4 inhibitors (e.g., diltiazem, ketoconazole)
10. Patient has a severe or fatal comorbid illness that will prevent improvement, or cannot complete follow-up due to the same, or cannot complete follow-up due to co-morbid non-fatal illness, non-residence in the city, or for any other known reason for which follow-up would be impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Composite rate of all-cause mortality, symptomatic intracranial bleeding, major extracranial bleeding | 180 days
  Symptomatic intracranial bleeding is defined as a new symptomatic intracranial hemorrhage OR worsening existing intracranial hemorrhage with a >33% change in hematoma volume, AND either an NIHSS score increase of 4 or more points, or a change in level of consciousness as per NIHSS item 1a, AND the clinical change is thought to be attributable to the hemorrhage.
  Major extracranial bleeding is defined as bleeding in a critical area or organ, including intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a drop in hemoglobin by 20 g/L or more, leading to transfusion of 2 or more units of whole blood or red cells.

SECONDARY OUTCOMES:
All-cause mortality | 180 days
  Death from any cause
Symptomatic intracranial bleeding | 180 days
  Symptomatic intracranial bleeding is defined as a new symptomatic intracranial hemorrhage OR worsening existing intracranial hemorrhage with a >33% change in hematoma volume, AND either an NIHSS score increase of 4 or more points, or a change in level of consciousness as per NIHSS item 1a, AND the clinical change is thought to be attributable to the hemorrhage.
Major extracranial bleeding | 180 days
  Major extracranial bleeding is defined as bleeding in a critical area or organ, including intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a drop in hemoglobin by 20 g/L or more, leading to transfusion of 2 or more units of whole blood or red cells.
Recurrent venous thromboembolism | 180 days or end of anticoagulation, whichever is sooner
  any thrombosis at a new site including cerebral venous thrombosis in a separate localization from index event
Major bleeding or clinically relevant non-major bleeding | 180 days or end of anticoagulation, whichever is sooner
  A clinically relevant minor bleed is an acute or subacute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of: (a) a hospital admission for bleeding, or (b) a physician guided medical or surgical treatment for bleeding, or (c) a change in antithrombotic therapy (including interruption or discontinuation or study drug)
Partial or complete recanalization | 180 or 365 days
  Partial or complete recanalization between baseline and last study venogram
Functional independence | 365 days
  modified Rankin Scale 0-1
Reduced functional dependence | 365 days
  shift of one or more modified Rankin Scale categories to reduced functional dependence
Health care resource utilization | 365 days
  Cost in Canadian dollars of number of hospitalizations (length of stay, critical care unit use), emergency room visits, unscheduled outpatient consultations, postacute care (including home care, rehabilitation stays or long-term care)
Population Health Questionnaire (PHQ)-9 score | 365 days
  Change in PHQ-9 score between baseline and end of study
EuroQOL 5-Dimensions (EQ-5D) score | 365 days
  Change in EQ-5D score between baseline and end of study
Fatigue Assessment score | 365 days
  Change in fatigue assessment score between baseline and end of study
Headache Impact Test - 6 score | 365 days
  Change in Headache Impact Test - 6 score between baseline and Day 180 (score = 36-78, where a higher score indicates a worse outcome)
Montreal Cognitive Assessment score | 365 days
  Change in performance on the Montreal Cognitive Assessment between baseline and end of study (score = 0-30, where a higher score indicates a better outcome)
National Institutes of Health toolbox - Cognitive battery score | 365 days
  Change in performance on the cognitive battery of the National Institutes of Health toolbox between baseline and end of study (where a higher score indicates a better outcome)
Boston cookie theft picture description task | 365 days
  Change in spontaneous speech between baseline and end of study. Components of spontaneous speech include lexical features (part-of-speech, word types and frequencies), syntactic complexity, grammaticality, fluency, vocabulary richness, and acoustic features.

CONTACTS AND LOCATIONS:
Overall Officials: Thalia S Field, MD FRCPC, Principal Investigator — University of British Columbia
Locations (11):
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the SECRET Trial, a public use database will be prepared by stripping any and all personal identifiers. The public use database, consisting of several data files, should contain: (1) baseline and demographic characteristics; (2) outcomes assessments; (3) CT/MRI data; (4) concomitant medications and procedures; and (5) adverse events. Each data file is made available as a formatted SAS dataset or other electronic format. The data files are distributed along with the data dictionary and a brief instruction ("Readme") file. These data files will be made available to the public only after all major manuscripts (including secondary analysis papers) of the Trial are accepted for publication in peer-reviewed journals.

REFERENCES:
- [Derived] Field TS, Dizonno V, Almekhlafi MA, Bala F, Alhabli I, Wong H, Norena M, Villaluna MK, King-Azote P, Ratnaweera N, Mancini S, Van Gaal SC, Wilson LK, Graham BR, Sposato LA, Blacquiere D, Dewar BM, Boulos MI, Buck BH, Odier C, Perera KS, Pikula A, Tkach A, Medvedev G, Canfield C, Mortenson WB, Nadeau JO, Alshimemeri S, Benavente OR, Demchuk AM, Dowlatshahi D, Lanthier S, Lee AYY, Mandzia J, Suryanarayan D, Weitz JI, Hill MD; SECRET Investigators. Study of Rivaroxaban for Cerebral Venous Thrombosis: A Randomized Controlled Feasibility Trial Comparing Anticoagulation With Rivaroxaban to Standard-of-Care in Symptomatic Cerebral Venous Thrombosis. Stroke. 2023 Nov;54(11):2724-2736. doi: 10.1161/STROKEAHA.123.044113. Epub 2023 Sep 7. PMID 37675613